CLINICAL TRIAL: NCT06199505
Title: A Phase II Trial Comparing Efficacy and Safety of GZR101 and Insulin Degludec/Insulin Aspart in Type 2 Diabetes Inadequately Controlled on Oral Antidiabetic Drug (OAD) Therapy or OAD Therapy in Combination with Insulin
Brief Title: A Trial Comparing Efficacy and Safety of GZR101 and IDegAsp in Insulin Naïve or Insulin Treated Subjects with T2DM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gan and Lee Pharmaceuticals, USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GL-GZR-CH2006
Record Dates: First submitted 2023-12-28; First posted 2024-01-10 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2023-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GZR101 (Experimental): GZR101 injection s.c., once daily, treat-to-target dose
  Interventions: Drug: GZR101
- insulin degludec/insulin aspart, (Active Comparator): insulin degludec/insulin aspart injection s.c., once or twice daily, treat-to-target dose
  Interventions: Drug: insulin degledec/insulin aspart

INTERVENTIONS:
Drug: GZR101 — Once daily
  Arms: GZR101
Drug: insulin degledec/insulin aspart — Once daily or twice daily
  Arms: insulin degludec/insulin aspart,

SUMMARY:
This trial is conducted in China. The aim of the trial is to compare the efficacy and safety of GZR101 and insulin degludec/insulin aspart in insulin naïve or insulin treated subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-75 years (both inclusive) at the time of signing informed consent.
* BMI = 18.5-35 kg/m2 (inclusive) at screening.
* Diagnosed with type 2 diabetes mellitus for ≥ 6 months.
* 7.0% ≤ HbA1c ≤ 11.0% at screening.

Exclusion Criteria:

* Women in pregnancy or lactation.
* Subjects with any malignancy diagnosed prior to screening or documented history of malignancy.
* Those with the following diseases within 6 months prior to screening: diabetic ketoacidosis, diabetic lactic acidosis, or hyperosmolar nonketotic diabetic coma.
* Subjects experiencing serious hypoglycaemic events (Level 3 hypoglycaemia) within 3 months prior to screening.
* Subjects with with history of acute heart failure or having been hospitalized for coronary heart disease, myocardial infarction, unstable angina, or stroke within 6 months prior to screening.
* Known or suspected hypersensitivity to trial product(s).
* Participation in a clinical study of another study drug within 1 month prior to randomization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | Baseline to week 16
  Change from baseline in HbA1c (Glycosylated Haemoglobin) after 16 weeks of treatment

SECONDARY OUTCOMES:
Change in Fasting Plasma Glucose (FPG) | Baseline to Week 16
  Change from baseline in fasting plasma glucose (FPG) after 16 weeks of treatment
The total daily dose of GZR101 and Insulin Degludec/Insulin Aspart at Week 16 | Week 16
  The total daily dose of GZR101 and the total daily dose of Insulin Degludec/Insulin Aspart at week 16 are presented.
Incidence and Rate of hypoglycemia Events | Baseline to Week 16
  Hypoglycaemia alert value (level 1) was defined as episodes that were sufficiently low for treatment with fast-acting carbohydrate and dose adjustment of glucose-lowering therapy with plasma glucose value of equal to or above (>=) 3.0 and less than (<) 3.9 mmol/L (>= 54 and < 70 mg/dL) confirmed by BG meter. Clinically significant hypoglycaemic episodes (level 2) were defined as episodes that were sufficiently low to indicate serious, clinically important hypoglycaemia with plasma glucose value of less than (<) 3.0 mmol/L (54 mg/dL). Severe hypoglycaemic episodes (level 3) were defined as episodes that were associated with severe cognitive impairment requiring external assistance for recovery. Severe hypoglycaemic episodes (level 3) were defined as episodes that were associated with severe cognitive impairment requiring external assistance for recovery.
Incidence and Rate of Treatment-emergent AE/SAEs | Baseline to Week 16
  A TEAE was defined as an event that had onset date (or increase in severity) during the on-treatment observation period.
Change from baseline in ADA and Nab | Baseline to Week 16
  Samples from the GZR101 arm of the study were analysed for anti-drug antibodies.

OTHER OUTCOMES:
Change from Baseline in Body Weight | Baseline to Week 16
  Change in body weight from baseline to week 16 is presented.

CONTACTS AND LOCATIONS:
Overall Officials: Chunyue Hao, PhD, Study Director — Gan & Lee Pharmaceuticals.
Locations (1):
- Gan & Lee Pharmaceuticals Co., Ltd, Beijing, Beijing Municipality, China